CLINICAL TRIAL: NCT03986372
Title: The Effect of Multiple Injection of Platlet-rich Plasma in Chronic Patellar Tendinopathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201900117A3
Record Dates: First submitted 2019-06-09; First posted 2019-06-14 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-08

CONDITIONS: Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP injection, once (Experimental): PRP injection, once
  Interventions: Biological: Platlet-rich plasma
- PRP injection, twice (Experimental): PRP injection, twice, 2 weeks apart
  Interventions: Biological: Platlet-rich plasma
- PRP injection, 3 times (Experimental): PRP injection, 3 times, 2 weeks apart
  Interventions: Biological: Platlet-rich plasma

INTERVENTIONS:
Biological: Platlet-rich plasma — Multiple Platlet-rich plasma injection.

SUMMARY:
According to previous studies, the effect of PRP to patellar tendinopathy could last longer. However, the type, concentration, time and frequent of injection are still debated。 This study is to understand the effect of multiple injection of platlet-rich plasma in chronic patellar tendinopathy and to analyze the relation between efficacy of PRP and the growth factor in PRP.

DETAILED DESCRIPTION:
Patellar tendinopathy, also known as jumper's knee，is clinically common characterised by anterior knee pain, activity-related pain、local tenderness over inferior pole of patella. The discomfort can result in decreasing athletic performance and be one of the most challenge for sports medicine doctor.

The patellar tendon suffer from repetitive microtrauma，result in reactive patellar tendinopathy. The overload tendon combining with risk factors of patellar tendinopathy will not recover timely and progress to chronic patellar tendinopathy. Hence, to reverse the progression is our aim.

According to previous studies, several nonsurgical treatment options have been proposed such as medication, eccentric exercise, corticosteroid injection, shockwave and platelet-rich plasma (PRP). Among all the options, the effect of PRP could last longer. However, the type, concentration, time and frequent of injection are still debated。Moreover, there is no study about the relationship between efficacy and the ratio and concentration of growth factor in the PRP.

The aim of this study is to understand (1) The effect of multiple injection of platlet-rich plasma in chronic patellar tendinopathy. (2) The effect of leukocyte-rich PRP in chronic patellar tendinopathy (3) Analyze the relation between efficacy of PRP and the growth factor in PRP.

ELIGIBILITY:
Inclusion Criteria:

Chronic patellar tendinopathy

Exclusion Criteria:

1. Corticosteroid injections within 12 months
2. Previous knee surgery
3. Any confounding diagnosis to the knee joint
4. Arthritis
5. Rheumatoid arthritis
6. Diabetes
7. Infections of knee joint
8. NSAIDs in the 10 days before the procedure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Victorian Institute of Sport Assessment (VISA-P) score to 36 weeks | 36 weeks
  Clinical evaluation for patellar tendinopathy minimum score: 0(worse outcome) maximum score: 100(better outcome)
Change from baseline modified Blazina Scale to 36 weeks | 36 weeks
  Clinical evaluation for patellar tendinopathy Stage 0 - No pain Stage 1 - Pain only after intense sports activity; no undue functional impairment Stage 2 - Pain at the beginning and after sports activity; still able to perform at a satisfactory level Stage 3 - Pain during sports activity; increasing difficulty in performing at a satisfactory level Stage 4 - Pain during sports activity; unable to participate in sport at a satisfactory level Stage 5 - Pain during daily activity; unable to participate in sport at any level
Change from baseline thickness of patellar tendon to 36 weeks | 36 weeks
  Sonographic evaluation for patellar tendinopathy to measure the thickness of proximal patellar tendon.
Change from baseline Visual analogue score(VAS) to 36 weeks | 36 weeks
  evaluation for pain(minimal score:0, maximal score:10)

SECONDARY OUTCOMES:
Correlation between Platlet derived growth factor (PDGF) and VISA-P score | 36 weeks
  Aim: To find the relationship between treatment effect(VISA-P score) and concentration of growth factor(PDGF)
Correlation between Transforming growth factor beta 1 (TGF beta 1) and VISA-P score | 36 weeks
  Aim: To find the relationship between treatment effect(VISA-P score) and concentration of growth factor(TGF beta 1)
Correlation between Epithelial growth factor (EGF) and VISA-P score | 36 weeks
  Aim: To find the relationship between treatment effect(VISA-P score) and concentration of growth factor(EGF)
Change from baseline Victorian Institute of Sport Assessment (VISA) score to 104 weeks | 104 weeks
  To evaluate the longterm effect of multiple PRP injection

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyuan Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No